CLINICAL TRIAL: NCT00478751
Title: Impact of Long Wavelength UVA and Visible Light on Melanocompetent Skin
Brief Title: Impact of Long Wavelength Ultraviolet (UVA) and Visible Light on Melanocompetent Skin
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Iltefat Hamzavi, Dermatologist, Henry Ford Health System
Other Study IDs: IRB4502
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Visible light, Long UVA,Pigmentation; Normal healthy volunteers with dark skin type.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* Determine the impact and the threshold of long wavelength UVA and visible light on immediate and delayed pigment production of melanocompetent individuals.
* The study basically wants to understand what types of light make us tan.

DETAILED DESCRIPTION:
1. Background:

   * A great deal is known about the impact of UVB and short wavelength UVA on pigmentation. Most sunscreens only protect against UVB and portions of UVA. However, it is not clear if other components of the spectrum of sunlight, not currently protected by sunscreens, are capable of eliciting pigmentation. Very little is known about the impact of long wavelength UVA and visible light on the time course to pigmentation, the quality of pigmentation and durations of this change in pigment if any. This has implications on the use of sunscreens to inhibit pigment production and the treatment of conditions that are aggravated by sun exposure such as melasma.
   * The impact of visible light (400-700 nm) on melanogenesis was studied by Porges et al in 1988 . The threshold dose for IPD with visible light was between 40 and 80 J/cm2, while the threshold dose for "persistent" pigmentation was greater than or equal to 80 J/cm2 (1).
2. Study objective:

   -To determine the impact of long wavelength UVA and visible light on immediate and delayed pigment production of melanocompetent individuals.
3. Study design:

   * Patient to serve as their own control. Patient must be melanocompetent (skin phototypes IV to VI) with no history of vitiligo, melasma or photosensitivity. The symmetric back or forearm will be used as a control of the irradiated area. Two phototherapy delivery system will be developed for the study: 1) A targeted visible light phototherapy device, 2) A targeted long wavelength UVA device.
   * Pigmentation will be assessed by visual exam, fluorescent and reflectance spectroscopy at 6 timepoints: immediately after irradiation, 30 minutes after exposure, 1 hour after exposure, 1 day after exposure, 1 week after exposure and 2 weeks after exposure.

ELIGIBILITY:
Inclusion Criteria:

For inclusion, the subject must:

1. Be at least 18 years old;
2. Be a healthy volunteer with Fitzpatrick Skin phototypes IV-VI based on the scale below:

   * Burns minimally, tans easily, and above average with each exposure
   * Rarely burns, tans easily and substantially
   * Never burns and tans profusely
3. Agree to abide by the Investigator's guidelines regarding photosensitizing drugs and photoprotection;
4. Be able to understand the requirements of the study, the risks involved, and be able to sign the informed consent form;
5. Agree to follow and undergo all study-related procedures.

Exclusion Criteria:

Subjects will be excluded if any of the following apply:

1. Women who are lactating, pregnant, or planning to become pregnant.
2. Patients with a recent history of vitiligo, melasma, and other disorders of pigmentation with the exception of post inflammatory hyperpigmentation.
3. Patients with a known history of photosensitivity disorders.
4. Photosensitizing medications may be continued throughout of the study at the discretion of the investigator (appendix A).
5. Patients with a known history of melanoma or non-melanoma skin cancers
6. Concomitant use of tanning beds.
7. Sun exposure of the irradiated or control areas.
8. Any reason the investigator feels the patient should not participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteer with Fitzpatrick Skin phototypes IV-VI.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iltefat H. Hamzavi, M.D., Principal Investigator — Department of Dermatology, Henry Ford Health System
Locations (1):
- Department of Dermatology, Henry Ford Medical Center, 3031 West Grand Boulevard,, Detroit, Michigan, United States

REFERENCES:
- [Background] Porges SB, Kaidbey KH, Grove GL. Quantification of visible light-induced melanogenesis in human skin. Photodermatol. 1988 Oct;5(5):197-200. PMID 3222167